CLINICAL TRIAL: NCT02002611
Title: Open Label, Randomized, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Lobeglitazone and Warfarin in Healthy Subjects
Brief Title: Drug-drug Interaction Study(Lobeglitazone, Warfarin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19DDI13016
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Lobeglitazone; Warfarin; Type 2 Diabetes Mellitus; Drug-Drug interaction; Phase 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lobeglitazone (Experimental): Subjects received Lobeglitazone 0.5 mg daily for 12 days in one period and in the other period, Subjects don't receive Lobeglitazone.
  Interventions: Drug: Lobeglitazone
- Warfarin (Experimental): Subjects received Warfarin 25 mg once at period 1 and 2.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Lobeglitazone
  Arms: Lobeglitazone
Drug: Warfarin
  Arms: Warfarin

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction between lobeglitazone and warfarin in healthy subjects.

DETAILED DESCRIPTION:
From day 1 to day 12, lobeglitazone 0.5mg is administered daily to Group 1 subjects during period 1. Then on day 5,warfarin 25mg is co-administered Group 1 subjects at period 1. After 10 day-break, warfarin 25mg is administered Group 1 subjects at period 2. On period 2, lobeglitazone is not administered.

Group 2 is administered in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male volunteer between 19 and 55 years old.
* BMI between 19 and 27.
* Signed the informed consent form prior to study participation.
* Able to participate in the entire trial

Exclusion Criteria:

* Clinically significant hepatic, renal, digestive system, respiratory system, endocrine system, nervous system, hematologic, cardiovascular system, tumor or have history of tumor
* Clinically significant hemorrhagic disease
* Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Have hypersensitivity reactions history for lobeglitazone, warfarin, excipient of IP or aspirin, antibiotics
* Medication which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products within 30 days prior to screening
* Participated in the other clinical trials and administrated IP within 60 days prior to screening
* Subject takes ethical drug or herbal medicine within 14 days, OTC within 7 days before screening
* Previously donate whole blood within 60 days or component blood within 30 days
* sit SBP < 90mmHg or sit SBP ≥ 140mmHg or sit DBP < 60mmHg or sit DBP ≥ 90mmHg
* A heavy alcohol consumer (alcohol > 140 g/week) or cannot stop drinking
* A heavy smoker (cigarette > 10 cigarettes per day) or cannot stop smoking
* A heavy caffeine consumer (more than 4cups per a day) or A heavy grapefruit consumer (more than 1cup per a day) or cannot stop having
* Positive for the Triage TOX drug on urine
* Positive for HIV antibody, HBsAg, HCV antibody test
* AST, ALT or Total bilirubin > UNL * 1.5
* Estimated GFR < normal limit
* INR, aPTT over the normal limit
* Clinically significant laboratory test result
* Clinically significant ECG
* An impossible one who participates in clinical trial by investigator's decision including other reason

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Assess AUC of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess Cmax of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess AUC of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess Cmax of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess AUC of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess Cmax of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h

SECONDARY OUTCOMES:
Assess tmax of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess t1/2 of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess CL/F of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess Vd/F of lobeglitazone | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24h
Assess tmax of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess t1/2 of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess CL/F of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess Vd/F of S-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess tmax of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess t1/2 of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess CL/F of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h
Assess Vd/F of R-warfarin | 0, 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168h

CONTACTS AND LOCATIONS:
Overall Officials: Jae Wook Ko, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea